CLINICAL TRIAL: NCT02800733
Title: The Effect of Saffron (Crocus Satious L.) in the Treatment of Mild to Moderate Generalized Anxiety Disorder: a Double Blind Randomized Controlled Trial
Brief Title: Effects of Saffron on Mild to Moderate Generalized Anxiety Disorder (GAD)
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: National Nutrition and Food Technology Institute (Other)
Responsible Party: Principal Investigator, Dr Azita Hekmatdoost, Dr Azita Hekmatdoost, National Nutrition and Food Technology Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 450/3654
Record Dates: First submitted 2016-06-11; First posted 2016-06-15 (Estimated); Last update posted 2016-06-15 (Estimated); Status verified 2016-06

CONDITIONS: Patients With Mild to Moderate GAD

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- saffron (Experimental): 450 mg of saffron capsule once a day for 6 weeks
  Interventions: Dietary Supplement: Saffron
- placebo (Placebo Comparator): placebo capsule once a day for 6 weeks
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: Saffron — 20 patients with mild to moderate GAD, diagnosed by Diagnostic and Statistical Manual of Mental Disorders-IѴ (DSM-IѴ) who receive sertraline will randomly receive saffron (450 mg) as an add-on therapy on daily bases for 6 weeks. Hamilton Anxiety Rating Scale (HAM-A) will use to assess the effect of treatment.
  Arms: saffron
Dietary Supplement: placebo — 20 patients with mild to moderate GAD who receive sertraline will receive placebo too
  Arms: placebo

SUMMARY:
anxiety disorder is one of the major public health problems worldwide. 25% of people experience anxiety disorders throughout life. Generalized anxiety disorder (GAD) is known as the most prevalent anxiety disorder. Saffron has previously approved as an effective adjuvant therapy in depression and might alleviate GAD symptoms.Since up to the best of our knowledge no human studies have assessed the therapeutic effect of saffron as an adjuvant therapy in GAD patients, Therefore, this study is planned to evaluateThe effect of saffron (Crocus satious L.) in the treatment of mild to moderate generalized anxiety disorder:

ELIGIBILITY:
Inclusion Criteria:

* Patients who diagnosed with GAD according to DSM-V criteria, Hamilton score of 18-25

Exclusion Criteria:

* pregnancy and lactation
* receiving antipsychotic medications in a month prior to the recruitment
* suffered from other psychological disorders (e.g. bipolar disorder, schizophrenia, mood disorders), and drug abuse

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-06; Primary Completion 2016-08 (Estimated); Study Completion 2016-09 (Estimated)

PRIMARY OUTCOMES:
Hamilton anxiety score | 6 weeks

IPD SHARING:
Plan to Share IPD: Undecided